CLINICAL TRIAL: NCT01891019
Title: Thalidomide in the Treatment of Chronic Plaque Psoriasis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-147; 21737
Record Dates: First submitted 2013-06-27; First posted 2013-07-02 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Psoriasis, Plaque-type
MeSH Terms: conditions — Psoriasis | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Thalidomide oral — Thalidomide will be administered nightly, with each subject taking 2 capsules totaling 100 milligrams for the initial two weeks of treatment, 3 capsules totaling 150 milligrams for week 2 to week 4, and 4 capsules totaling 200 milligrams for week 4 to end of treatment. The subjects will take the medication for 12 weeks.
  Other Names: Thalomid

SUMMARY:
The objective of this study is to obtain information on the effectiveness of thalidomide in psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 years of age or older.
* Stable or worsening psoriasis that involves 5% or greater of total body surface area (BSA) involvement with a minimum PASI score of 8.
* Moderate to severe plaque-type psoriasis, defined by a minimum score of 1 for each of erythema, scaling, and plaque thickness (using a 0 - 4 scale).
* Patients receiving systemic retinoids, prednisone, methotrexate, or cyclosporine should be on a stable dose at least 28 days prior to the first dose of thalidomide.
* Patients receiving topical treatments should be consistent with such treatments throughout the study.
* The ability and willingness to follow all study procedures, attend all scheduled visits, and successfully complete the study.
* The ability to understand and sign a written informed consent form, which must be obtained prior to treatment.
* The ability to understand, agree to, and comply with the requirements of the System for Thalidomide Education and Prescribing Safety (S.T.E.P.S.).**

(*Because of the known teratogenic effects of thalidomide and in an effort to prevent to the greatest extent possible any chance of fetal exposure to thalidomide, THALOMID(thalidomide) is approved for marketing only under a special restricted distribution program approved by the FDA. Under this program, the System for Thalidomide Education and Prescribing Safety (S.T.E.P.S.), only prescribers and pharmacists registered with the program are allowed to prescribe and dispense thalidomide (Zeldis JB et al. 1999). In addition, patients must be advised of, agree to, and comply with the requirements of the S.T.E.P.S. Program. To monitor patient compliance with the S.T.E.P.S. program, all patients must complete the S.T.E.P.S. program informed consent and participate in a mandatory and confidential surveillance registry.)

Exclusion Criteria:

* Unstable psoriasis
* Unable or unwilling to meet all criteria for contraception as required in STEPS.
* Known allergy to thalidomide.
* Known history of neuropathy.
* Abnormal laboratory test results that the investigator feels would compromise patient safety or evaluation of drug safety.
* The introduction of drugs for other medical conditions which are known to affect psoriasis (e.g., lithium, beta-adrenergic blockers, etc.) during the period 4 weeks prior to and during the study period.
* Use of any investigational therapy within the 4 weeks prior to the first dose of thalidomide.
* Expectation of exposure to strong sunlight during the course of the study (e.g. planned holiday in high sunlight area) or intention of sunbathing for prolonged periods of time during the course of the study.
* Current drug or alcohol abuse (drug screening not required).
* Medical conditions that preclude thalidomide therapy. Any other condition which, in the judgment of the investigator, would put the subject at unacceptable risk for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2003-04; Primary Completion 2005-09 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) Score | 12 weeks
  The change from Baseline to Week 12 (or end of treatment) in the composite score (PASI) of the signs of psoriasis (erythema, scaling, plaque thickness).

SECONDARY OUTCOMES:
Subject Global Assessment | 4 months
  Investigator and Subject Global Assessment of Response at Weeks 2, 4, 8, 12 (or end of treatment) and at Week 16 (follow-up).

OTHER OUTCOMES:
Pruritus Score | 12 week
  The change in pruritus score from Baseline to Week 12 (or end of treatment).
  The pruritus grading system (PGS) score for each patient was based on: distribution, frequency,severity of itch and quality of sleep. Each patient's itch grade is calculated as the sum of the individual scores as:
  Mild grade: if total score is between 0 and 5. Moderate grade: if total score is between 6 and 11. Severe grade: if total score is between 12 and 19.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Feldman, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Dermatology, Winston-Salem, North Carolina, United States